CLINICAL TRIAL: NCT06982586
Title: A Prospective, Single-Center, Single-Arm, Investigator-Initiated Exploratory Clinical Trial to Assess the Safety of Repetitive Transcranial Magnetic Stimulation for Children and Adolescents With Autism Spectrum Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle Investigator, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-02-028
Record Dates: First submitted 2025-05-11; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repetitive transcranial magnetic stimulation (Experimental): Repetitive transcranial magnetic stimulation
  Interventions: Device: Repetitive transcranial magentic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magentic stimulation — Low frequencey repetitive transcranial magentic stimulation

SUMMARY:
This is a prospective, single-center, single-arm, investigator-initiated exploratory clinical trial aimed at evaluating the safety and exploring the efficacy of a medical electromagnetic stimulator delivering low-frequency repetitive transcranial magnetic stimulation (rTMS) in children and adolescents with Autism Spectrum Disorder (ASD). ASD is a neurodevelopmental disorder characterized by deficits in social interaction and communication and restricted, repetitive behaviors. Despite increasing prevalence, effective treatment options remain limited, and the demand for non-invasive, safe interventions continues to grow.

In this study, a total of 18 participants aged 3 to 17 years with a clinical diagnosis of ASD will be enrolled. Participants will receive rTMS using a medically approved electromagnetic stimulator applied to the dorsolateral prefrontal cortex (DLPFC) - five sessions per week for two consecutive weeks (total of 10 sessions). The first 5 sessions will target the left DLPFC, and the remaining 5 will target the right DLPFC. Each session includes 18 trains of 10-second stimulations at 1Hz frequency with 20-second inter-train intervals. The stimulation intensity is set at 90% of the resting motor threshold (rMT), determined individually using motor evoked potential testing.

The primary objective of this trial is to assess the safety of low-frequency rTMS in this population, with adverse events such as seizures, headaches, dizziness, and mood changes monitored throughout the trial. Vital signs will also be checked before and after each session. Secondary objectives include exploratory evaluation of rTMS effects on sensory processing (SP), social communication (SCQ), autism severity (K-CARS), behavioral symptoms (CBCL), brain activity changes (fNIRS), and electrophysiological responses (EEG), assessed at baseline, immediately after intervention, and at 1- and 3-month follow-ups.

All participants will undergo baseline assessments including EEG, SP, SCQ, K-CARS, CBCL, fNIRS, and vital signs. These measures will be repeated after the final rTMS session, and again at 1 and 3 months post-intervention. The trial will be conducted at CHA Bundang Medical Center, led by Principal Investigator Professor Minyoung Kim, Department of Rehabilitation Medicine.

This exploratory study is designed to provide preliminary evidence for the safety of low-frequency rTMS in ASD and to gather pilot data on its potential therapeutic effects, which may support future randomized controlled trials and clinical applications.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 3 and 17 years at the time of enrollment
2. Clinically diagnosed with Autism Spectrum Disorder (ASD), including assessment using the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)
3. Currently receiving outpatient care for ASD at the Department of Rehabilitation Medicine, CHA Bundang Medical Center
4. The participant and their legal guardian have been fully informed of the study and have voluntarily provided written informed consent

Exclusion Criteria:

1. Diagnosed with a major neurological condition other than ASD
2. Epileptiform discharges detected on EEG screening requiring initiation or adjustment of antiepileptic medication
3. Diagnosed with other psychiatric disorders, such as schizophrenia or major depressive disorder
4. History of traumatic brain injury, brain tumor, or other significant brain conditions
5. Deemed unsuitable for participation by the principal investigator
6. Currently participating in another interventional clinical trial, or has participated in one within the past 30 days (excluding observational studies)
7. Any of the following contraindications to rTMS:

   * Implanted electronic medical devices (e.g., pacemaker)
   * Presence of metal implants in the skull
   * Skin lesions at the stimulation site
   * History of epilepsy
   * Cervical spine pain or musculoskeletal disorders
   * Pregnancy or currently breastfeeding

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Characteristics of Adverse Events Related to rTMS Treatment in Children and Adolescents with Autism Spectrum Disorder | From baseline (Day 1) through end of follow-up at 3 months after the final rTMS session (approximately 90 days)
  This outcome measure assesses the safety of applying low-frequency repetitive transcranial magnetic stimulation (rTMS) using a medical electromagnetic stimulator in children and adolescents diagnosed with Autism Spectrum Disorder (ASD). All adverse events (AEs), including seizures, syncope, headaches, local pain, hearing problems, dizziness, mood disturbances, or other subjective discomforts, will be recorded during the study period. The severity and relationship of AEs to the intervention will be classified using standardized criteria (e.g., CTCAE v5.0). Vital signs will be monitored before and after each session to support safety evaluation.

SECONDARY OUTCOMES:
Change in Sensory Profile (SP) Score | Baseline (Day 1), Post-intervention (Day 12), 1-month follow-up (Day ~30), 3-month follow-up (Day ~90)
  This outcome evaluates changes in sensory processing characteristics before and after the rTMS intervention using the Sensory Profile questionnaire. The aim is to explore whether low-frequency rTMS modulates sensory regulation in children and adolescents with ASD.
Change in Social Communication Questionnaire (SCQ) Score | Baseline (Day 1), Post-intervention (Day 12), 1-month follow-up (Day ~30), 3-month follow-up (Day ~90)
  This measure assesses changes in social communication behaviors following rTMS intervention. The SCQ evaluates communication skills and social functioning relevant to autism characteristics.
Change in Korean-Childhood Autism Rating Scale, 2nd Edition (K-CARS-2) Score | Baseline (Day 1), Post-intervention (Day 12), 3-month follow-up (Day ~90)
  This outcome examines changes in autism severity by comparing K-CARS-2 scores across time points, investigating whether rTMS reduces core ASD symptoms.
Change in Child Behavior Checklist (CBCL) Score | Baseline (Day 1), Post-intervention (Day 12), 1-month follow-up (Day ~30), 3-month follow-up (Day ~90)
  This measure explores changes in emotional and behavioral functioning post-rTMS, using the CBCL, a parent-reported instrument capturing internalizing and externalizing problems.
Change in Functional Near-Infrared Spectroscopy (fNIRS) Signals | Baseline (Day 1), 3-month follow-up (Day ~90)
  This neuroimaging-based outcome assesses changes in cortical hemodynamic responses during cognitive and social tasks using fNIRS, particularly targeting the prefrontal cortex before and after rTMS.
Change in Electroencephalography (EEG) Patterns | Baseline (Day 1), 3-month follow-up (Day ~90)
  Electroencephalography (EEG) will be recorded using a standard 10-20 electrode placement system. The power spectral density (PSD) will be computed for the following frequency bands:
  * Delta (1-4 Hz)
  * Theta (4-8 Hz)
  * Alpha (8-13 Hz)
  * Beta (13-30 Hz) Mean absolute and relative band power within these bands will be calculated for frontal, central, and parietal electrodes. Changes from baseline to post-intervention and follow-up periods will be analyzed to assess neuromodulatory effects of rTMS. Artifacts will be removed using independent component analysis (ICA).

IPD SHARING:
Plan to Share IPD: No